CLINICAL TRIAL: NCT03136640
Title: Multicenter Safety, Feasibility and Pharmacokinetic Phase I Trial of ModraDoc006/r in Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: ModraDoc006/r in Metastatic Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Modra Pharmaceuticals (Industry)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M17DOC
Record Dates: First submitted 2017-04-25; First posted 2017-05-02 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2020-12

CONDITIONS: Castration-resistant Prostate Cancer

STUDY DESIGN:
Intervention Model Description: Three patients will start at the starting dose level. If none of these patients experiences a DLT, another three patients will be added at the same dose level. The dose will be escalated or de-escalated based on safety and pharmacokinetic parameters. The recommended dose level, defined as the maximum tolerated dose (MTD) of docetaxel (as ModraDoc006 10 mg tablets) that can safely be administered in combination with ritonavir to patients with metastatic castration-resistant prostate cancer in a bi-daily weekly schedule without interruption and results in an adequate systemic exposure to docetaxel, will be expanded to at least 20 for toxicity evaluable patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ModraDoc006/r (Experimental): Weekly ModraDoc006/r treatment as ModraDoc006 (oral docetaxel) 10mg tablets combined with ritonavir 100mg tablets
  Interventions: Drug: ModraDoc006/r

INTERVENTIONS:
Drug: ModraDoc006/r — Treatment with weekly ModraDoc006 (oral docetaxel) 10mg tablets in combination with ritonavir 100mg tablets
  Other Names: oral docetaxel formulation

SUMMARY:
This is a safety, feasibility and pharmacokinetic study to confirm that the recommended safe dose and schedule of ModraDoc006/r (oral docetaxel with ritonavir) as determined in a previous phase I study is also safe and feasible in the target population of patients with CRPC.

DETAILED DESCRIPTION:
This is a safety, feasibility and pharmacokinetic phase II study to evaluate treatment with ModraDoc006/r (oral docetaxel with ritonavir) in chemotherapy naïve patients with castration-resistant metastatic prostate cancer for whom treatment with intravenous docetaxel is indicated. The primary objective of this study is to determine the recommended dose determined as the maximum tolerated dose (MTD) of docetaxel (as ModraDoc006 10 mg tablets) that can safely be administered in combination with ritonavir to patients with metastatic castration-resistant prostate cancer in a bi-daily weekly schedule without interruption and results in an adequate systemic exposure to docetaxel. On a predefined day of the first and every subsequent week, the patient will receive oral docetaxel (as ModraDoc006 10 mg tablets). This regime will be continued weekly (intake around the same time) until completion of the study, progressive disease or until adverse events, which require dose modification or discontinuation of therapy, are observed.

A dose escalation design will be used to determine the recommended dose of ModraDoc006 in combination with ritonavir that is safe and feasible and provides an adequate systemic docetaxel exposure in the target population of the projected pivotal study in patients with CRPC. Three castration-resistant metastatic prostate cancer (CRPC) patients will be assigned to the starting dose level 1A of 30-20 mg ModraDoc006 in a bi-daily weekly schedule, each intake of ModraDoc006 will be combined with 200 mg ritonavir. If no more than one DLT has occurred during the first four weeks of treatment on dose level 1A (30-20 mg ModraDoc006 and bi-daily ritonavir 200 mg) and the pharmacokinetic results are favorable, than three additional patients will be added to this dose level. If no more than 1 DLT in these first 6 patients has occurred, this will be the recommended dose and this dose level will be expanded until a total of 20 for toxicity evaluable patients have been treated on this dose level.

If 2 DLTs have occurred directly in the first 3 patients or in the first 6 patients (after the previous described addition of 3 patients), during the first four weeks of treatment on dose level 1A (30-20 mg ModraDoc006 and bi-daily 200 mg ritonavir) and the pharmacokinetic results are favorable, the dose may be de-escalated to the next lower dose-level, depending on the pharmacokinetic results and the study schedule will start again from the beginning.

If no more than one DLT has occurred in the first 6 patients during the first four weeks of treatment on dose level 1A and the pharmacokinetic results are not favorable, than the dose will be escalated depending on the pharmacokinetic results and the study schedule will start again from the beginning.

If two or more DLTs have occurred in the first 6 patients during the first four weeks of treatment on dose level 1A and the pharmacokinetic results are not favorable, the dose will be altered according to the type of DLT.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological proven castration-resistant metastatic prostate cancer with an indication for systemic treatment with intravenous docetaxel at the discretion of the physician
2. Progressive disease defined as biochemical and/or radiological progression according to the Prostate Cancer Working group 3 recommendations.
3. Disease evaluable for biochemical and/or radiological response (in case disease is measurable the RECIST 1.1 criteria and the guidelines for measurement of bone lesions according to the Prostate Cancer Clinical Trials Working Group 3 will be applied, as described in "Efficacy assessment").
4. Chemotherapy naïve patients. Prior treatment with abiraterone or enzalutamide as first line therapy is allowed. In case of use of enzalutamide, this should be stopped 2 weeks before the first ModraDoc006/r intake. For patients that have used enzalutamide, altered pharmacokinetic sampling should be done, as described at 'Pharmacokinetics and Circulating Tumour Cell measurements"
5. Castrate levels of testosterone, defined as ≤ 50 ng/dL (or ≤ 0.50 ng/mL or 1.73 nmol/L)
6. Age equal or above 18 years
7. Adequate haematological, renal and hepatic functions
8. WHO performance status of 0-2
9. Life expectancy above 3 months allowing adequate follow up of toxicity evaluation and antitumor activity;
10. Able and willing to swallow oral medication
11. Able and willing to undergo blood sampling
12. Able and willing to give written informed consent

Exclusion Criteria:

1. Any treatment with investigational drugs, chemotherapy or immunotherapy within 28 days prior to receiving the first dose of investigational treatment. Palliative radiotherapy is allowed before and during the study as long as this is scheduled outside the DLT-period (first 28 days) and at least 4 days after intake of study medication and no intestinal toxicity is expected from the radiotherapy.
2. Patients with symptomatic brain metastases. Patients previously treated or untreated for these conditions that are asymptomatic in the absence of corticosteroid and anticonvulsant therapy for at least 6 weeks are allowed to enroll. Radiotherapy for brain metastasis must have been completed at least 6 weeks prior to start of study treatment. Brain metastasis must be stable with verification by imaging (e.g. brain MRI or CT completed at screening, demonstrating no current evidence of progressive brain metastases). Patients are not permitted to receive anti-epileptic drugs or corticosteroid treatment indicated for brain metastasis. Patients with a history of leptomeningeal metastases are not eligible.
3. Unreliable contraceptive methods. Men enrolled in this trial must agree to use a reliable contraceptive method throughout the study (adequate contraceptive methods are: condom, sterilization, other barrier contraceptive measures preferably in combination with condoms)
4. Unresolved (> grade 1) toxicities of previous therapy, excluding alopecia.
5. Uncontrolled infectious disease or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients;
6. Patients with a known history of hepatitis B or C;
7. Bowel obstructions or motility disorders that may influence the resorption of drugs as judged by the treating physician
8. Concomitant use of MDR and CYP3A modulating drugs such as Ca+- entry blockers (verapamil, dihydropyridines), cyclosporine, quinidine, tamoxifen, megestrol and grapefruit juice, concomitant use of HIV medications, other protease inhibitors, (non) nucleoside analogues, or St. John's wort.
9. Use of Bicalutamide within 14 days prior to receiving the first dose of investigational treatment
10. Patients with known alcoholism, drug addiction and/or psychiatric of physiological condition which in the opinion of the investigator would impair study compliance; Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
11. Legal incapacity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of ModraDoc006/r treatment | Safety and tolerance will be evaluated using the CTCAEv4.03 grading system, dose limiting toxicities will be evaluated during the first 4 weeks of treatment
  The maximum tolerated dose (MTD) of docetaxel (as ModraDoc006 10 mg tablets) that can safely be administered in combination with ritonavir to patients with metastatic castration-resistant prostate cancer in a bi-daily weekly schedule without interruption

SECONDARY OUTCOMES:
The AUC of docetaxel (area under the curve) | Pharmacokinetic sampling during week 1 and week 2, 0-48 hrs after administration (i.e. the first 2 treatment cycles)
  The AUC of docetaxel given as bi-daily ModraDoc006 10 mg tablets in combination with ritonavir
The cMax (peak concentration) of docetaxel | Pharmacokinetic sampling during week 1 and week 2, 0-48 hrs after administration (i.e. the first 2 treatment cycles)
  The cMax (peak concentration) of docetaxel given as bi-daily ModraDoc006 10 mg tablets in combination with ritonavir
The hematological and non-hematological toxicity profile of oral docetaxel in combination with ritonavir | Safety and tolerance will be evaluated during the complete study treatment until 28 days after the last intake, using the CTCAEv4.03 grading system]
  The number of CTCAE v.4.03 grade 3-4 toxicities during treatment with ModraDoc006/r
The preliminary anti-tumor activity of the oral docetaxel formulation | PSA and radiological evaluation every 6 weeks, up to 30 weeks
  PSA response, radiological response of visceral and nodal lesions according to RECIST 1.1, progression of bone lesions according to Prostate Cancer Working Group 3 criteria
The dose limiting toxicities (DLT) of ModraDoc006/r treatment | First 4 weeks of treatment
  Determine dose limiting toxicities (DLT) and recommended dose (RD) of ModraDoc006/r that can safely be administered to patients with metastatic castration-resistant prostate cancer in a bi-daily weekly schedule

CONTACTS AND LOCATIONS:
Overall Officials: Andre Bergman, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (4):
- Netherlands (4):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vermunt MAC, van der Heijden LT, Hendrikx JJMA, Schinkel AH, de Weger VA, van der Putten E, van Triest B, Bergman AM, Beijnen JH. Pharmacokinetics of docetaxel and ritonavir after oral administration of ModraDoc006/r in patients with prostate cancer versus patients with other advanced solid tumours. Cancer Chemother Pharmacol. 2021 Jun;87(6):855-869. doi: 10.1007/s00280-021-04259-5. Epub 2021 Mar 20. PMID 33744986